CLINICAL TRIAL: NCT05028244
Title: Systematic Ultrasound Screening for Lower Extremity Deep Vein Thrombosis in ICU Patients With Severe COVID-19: a Randomized Clinical Trial.
Brief Title: Evaluation of Serial Ultrasound Screening in ICU COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P/R(AG)176/2021
Record Dates: First submitted 2021-08-30; First posted 2021-08-31 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Deep Vein Thrombosis; Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Acute Bronchitis; COVID-19 Lower Respiratory Infection; Pulmonary Embolism
Keywords: covid19; pulmonary embolism; intensive care unit; deep venous thrombosis
MeSH Terms: conditions — Venous Thrombosis; COVID-19; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: The selected patients undergo an ultrasound of lower extremity to discard previous thrombosis episodes. Then they are randomized to an intervention group (serial screening of deep venous thrombosis in lower extremity 2 times per week) or control group (no other exploration or interventions are made).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Selected patients undergo lower extremity ultrasound for diagnosis of deep vein thrombosis 2 times per week (Mondays and Thursdays) in a period of 3 weeks (21 days) of follow up
  Interventions: Diagnostic Test: venous ultrasound of lower extremity
- control group (No Intervention): This group only undergo the first ultrasound assessment to discard previous thrombosis not detected during hospitalisation or ambulatory

INTERVENTIONS:
Diagnostic Test: venous ultrasound of lower extremity — Patients are explored for deep vein thrombosis in femoral-popliteal and distal veins of the legs with ultrasound compression and doppler flow evaluation
  Arms: Intervention group

SUMMARY:
This clinical trial is designed to evaluate if the periodic screening for deep venous thrombosis by ultrasound of lower extremity in patients with intensive care unit (ICU) patients with COVID 19 impacts on mortality, ICU stay and total length of stay in the hospital, along with other outcomes.

DETAILED DESCRIPTION:
Background: COVID-19 has a high incidence of venous thromboembolic disease (VTE), especially pulmonary thromboembolism (PE) and deep vein thrombosis (DVT), with an even higher incidence in patients admitted to the intensive care unit (ICU). The presentation of these events is related to an increase in mortality and the mean stay in the ICU. The impact of systematic screening for asymptomatic lower extremity DVT in these patients has not been studied, so we propose to carry out a clinical trial to assess its impact in these patients.

Hypothesis: Serial DVT screening in patients admitted to the ICU for COVID-19 does not improve survival, mean stay, or the incidence of symptomatic VTE.

Objective: To study whether DVT screening in these patients has an impact on the incidence of symptomatic VTE, mortality and average stay in the ICU.

Methods: Non-blind randomized clinical trial on all patients aged 18 years or older admitted to the ICU for COVID-19 with less than 72 hours elapsed since their admission to the unit. Patients with DVT or PE will be excluded at the time of recruitment (all patients will be ruled out by routine ultrasound and computed tomography angiography (CT Angiography)); Pregnant patients, patients with a previous diagnosis of DVT or PE, and patients undergoing extracorporeal membrane oxygenation (ECMO) will also be excluded. Patients will be randomized into two arms at the time of inclusion: the screened group (Group 1) and the non-screened group (Group 2). Group 1: patients who will be treated according to the usual ICU protocol and, additionally, will undergo serial ultrasounds of the lower extremities twice a week (Monday and Thursday). Group 2: they will be treated according to the usual ICU protocol and no screening examinations will be performed. Patients will be followed until discharge from the ICU or death and up to a maximum of 3 weeks. The incidence of symptomatic VTE will be assessed, as well as all-cause mortality and days of stay in the ICU. Clinical and laboratory variables will be collected from each patient for subsequent statistical analysis.

Relevance: The thrombotic complications of COVID-19 are well described, as well as their high incidence in critically ill patients. This work aims to clarify the current doubts about the need for systematic DVT screening in these patients. If our hypothesis is verified, a limited resource such as ultrasound of the lower limbs could be saved, as well as the use of the necessary protection materials and, most importantly, avoid unnecessary exposure of health personnel with the consequent risk that it represents for other professionals and patients.

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 patients in their first 72 hours of entering ICU

Exclusion Criteria:

* Pregnant patients
* Not COVID 19 confirmed patients by RCP
* Patients that are in Extracorporeal membrane oxygenation
* Patients with previous thrombotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Mortality | 21 days
  Patients that die in ICU during follow up
ICU Stay | 21 days
  Number of days staying in that unit during follow up
Symptomatic deep venous thrombosis | 21 days
  presence of confirmed deep vein thrombosis and presence of symptoms

SECONDARY OUTCOMES:
composite outcome | 21 days
  a composite outcome with poor outcome factors (symptomatic DVT, bleeding, ICU stay >21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Bellmunt Montoya, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wells PS, Anderson DR, Bormanis J, Guy F, Mitchell M, Gray L, Clement C, Robinson KS, Lewandowski B. Value of assessment of pretest probability of deep-vein thrombosis in clinical management. Lancet. 1997 Dec 20-27;350(9094):1795-8. doi: 10.1016/S0140-6736(97)08140-3. PMID 9428249
- [Background] Jenner WJ, Kanji R, Mirsadraee S, Gue YX, Price S, Prasad S, Gorog DA. Thrombotic complications in 2928 patients with COVID-19 treated in intensive care: a systematic review. J Thromb Thrombolysis. 2021 Apr;51(3):595-607. doi: 10.1007/s11239-021-02394-7. Epub 2021 Feb 14. PMID 33586113
- [Background] Mohamed MFH, Al-Shokri SD, Shunnar KM, Mohamed SF, Najim MS, Ibrahim SI, Elewa H, Abdalla LO, El-Bardissy A, Elshafei MN, Abubeker IY, Danjuma M, Dousa KM, Yassin MA. Prevalence of Venous Thromboembolism in Critically Ill COVID-19 Patients: Systematic Review and Meta-Analysis. Front Cardiovasc Med. 2021 Jan 8;7:598846. doi: 10.3389/fcvm.2020.598846. eCollection 2020. PMID 33585578
- [Background] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Background] Sebuhyan M, Mirailles R, Crichi B, Frere C, Bonnin P, Bergeron-Lafaurie A, Denis B, Liegeon G, Peyrony O, Farge D; Saint-Louis CORE (COVID-19 RESEARCH) group. How to screen and diagnose deep venous thrombosis (DVT) in patients hospitalized for or suspected of COVID-19 infection, outside the intensive care units. J Med Vasc. 2020 Dec;45(6):334-343. doi: 10.1016/j.jdmv.2020.08.002. Epub 2020 Sep 4. PMID 33248536
- [Background] Boonyawat K, Chantrathammachart P, Numthavaj P, Nanthatanti N, Phusanti S, Phuphuakrat A, Niparuck P, Angchaisuksiri P. Incidence of thromboembolism in patients with COVID-19: a systematic review and meta-analysis. Thromb J. 2020 Nov 23;18(1):34. doi: 10.1186/s12959-020-00248-5. PMID 33292258
- [Background] Jimenez D, Garcia-Sanchez A, Rali P, Muriel A, Bikdeli B, Ruiz-Artacho P, Le Mao R, Rodriguez C, Hunt BJ, Monreal M. Incidence of VTE and Bleeding Among Hospitalized Patients With Coronavirus Disease 2019: A Systematic Review and Meta-analysis. Chest. 2021 Mar;159(3):1182-1196. doi: 10.1016/j.chest.2020.11.005. Epub 2020 Nov 17. PMID 33217420
- [Background] Suh YJ, Hong H, Ohana M, Bompard F, Revel MP, Valle C, Gervaise A, Poissy J, Susen S, Hekimian G, Artifoni M, Periard D, Contou D, Delaloye J, Sanchez B, Fang C, Garzillo G, Robbie H, Yoon SH. Pulmonary Embolism and Deep Vein Thrombosis in COVID-19: A Systematic Review and Meta-Analysis. Radiology. 2021 Feb;298(2):E70-E80. doi: 10.1148/radiol.2020203557. Epub 2020 Dec 15. PMID 33320063
- [Background] Bohula EA, Berg DD, Lopes MS, Connors JM, Babar I, Barnett CF, Chaudhry SP, Chopra A, Ginete W, Ieong MH, Katz JN, Kim EY, Kuder JF, Mazza E, McLean D, Mosier JM, Moskowitz A, Murphy SA, O'Donoghue ML, Park JG, Prasad R, Ruff CT, Shahrour MN, Sinha SS, Wiviott SD, Van Diepen S, Zainea M, Baird-Zars V, Sabatine MS, Morrow DA; COVID-PACT Investigators. Anticoagulation and Antiplatelet Therapy for Prevention of Venous and Arterial Thrombotic Events in Critically Ill Patients With COVID-19: COVID-PACT. Circulation. 2022 Nov;146(18):1344-1356. doi: 10.1161/CIRCULATIONAHA.122.061533. Epub 2022 Aug 29. PMID 36036760
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers D, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Confirmation of the high cumulative incidence of thrombotic complications in critically ill ICU patients with COVID-19: An updated analysis. Thromb Res. 2020 Jul;191:148-150. doi: 10.1016/j.thromres.2020.04.041. Epub 2020 Apr 30. PMID 32381264
- [Background] Gil-Sala D, Riera C, Garcia-Reyes M, Rodriguez M, Marrero CE, Martinez L, Gil M, Ruiz-Rodriguez JC, Ferrer R, DE Nadal M, Suito-Alcantara MA, Llagostera S, Bellmunt-Montoya S. Mortality and bleeding complications of COVID-19 critically ill patients with venous thromboembolism. Int Angiol. 2022 Feb;41(1):1-8. doi: 10.23736/S0392-9590.21.04704-0. Epub 2021 Nov 9. PMID 34751541
- [Background] Mansory EM, Srigunapalan S, Lazo-Langner A. Venous Thromboembolism in Hospitalized Critical and Noncritical COVID-19 Patients: A Systematic Review and Meta-analysis. TH Open. 2021 Jul 6;5(3):e286-e294. doi: 10.1055/s-0041-1730967. eCollection 2021 Jul. PMID 34240001
- [Background] Xiao D, Tang F, Chen L, Gao H, Li X. Cumulative Evidence for the Association of Thrombosis and the Prognosis of COVID-19: Systematic Review and Meta-Analysis. Front Cardiovasc Med. 2022 Jan 25;8:819318. doi: 10.3389/fcvm.2021.819318. eCollection 2021. PMID 35146009
- [Background] Mazzaccaro D, Giannetta M, Fancoli F, Milani V, Modafferi A, Malacrida G, Righini P, Marrocco-Trischitta MM, Nano G. COVID and venous thrombosis: systematic review of literature. J Cardiovasc Surg (Torino). 2021 Dec;62(6):548-557. doi: 10.23736/S0021-9509.21.12022-1. Epub 2021 Sep 14. PMID 34520137
- [Background] Kollias A, Kyriakoulis KG, Lagou S, Kontopantelis E, Stergiou GS, Syrigos K. Venous thromboembolism in COVID-19: A systematic review and meta-analysis. Vasc Med. 2021 Aug;26(4):415-425. doi: 10.1177/1358863X21995566. Epub 2021 Apr 4. PMID 33818197
- [Background] Tufano A, Rendina D, Abate V, Casoria A, Marra A, Buonanno P, Galletti F, Di Minno G, Servillo G, Vargas M. Venous Thromboembolism in COVID-19 Compared to Non-COVID-19 Cohorts: A Systematic Review with Meta-Analysis. J Clin Med. 2021 Oct 25;10(21):4925. doi: 10.3390/jcm10214925. PMID 34768445
- [Background] Malas MB, Naazie IN, Elsayed N, Mathlouthi A, Marmor R, Clary B. Thromboembolism risk of COVID-19 is high and associated with a higher risk of mortality: A systematic review and meta-analysis. EClinicalMedicine. 2020 Dec;29:100639. doi: 10.1016/j.eclinm.2020.100639. Epub 2020 Nov 20. PMID 33251499
- [Background] Zhang R, Ni L, Di X, Wang X, Ma B, Niu S, Liu C. Systematic review and meta-analysis of the prevalence of venous thromboembolic events in novel coronavirus disease-2019 patients. J Vasc Surg Venous Lymphat Disord. 2021 Mar;9(2):289-298.e5. doi: 10.1016/j.jvsv.2020.11.023. Epub 2020 Dec 9. PMID 33309903
- [Background] Reis S, Popp M, Schmid B, Stegemann M, Metzendorf MI, Kranke P, Meybohm P, Weibel S. Safety and Efficacy of Intermediate- and Therapeutic-Dose Anticoagulation for Hospitalised Patients with COVID-19: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Dec 23;11(1):57. doi: 10.3390/jcm11010057. PMID 35011804
- [Background] Moonla C, Sosothikul D, Chiasakul T, Rojnuckarin P, Uaprasert N. Anticoagulation and In-Hospital Mortality From Coronavirus Disease 2019: A Systematic Review and Meta-Analysis. Clin Appl Thromb Hemost. 2021 Jan-Dec;27:10760296211008999. doi: 10.1177/10760296211008999. PMID 33874753
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Cui S, Chen S, Li X, Liu S, Wang F. Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia. J Thromb Haemost. 2020 Jun;18(6):1421-1424. doi: 10.1111/jth.14830. Epub 2020 May 6. PMID 32271988
- [Background] Bellmunt-Montoya S, Riera C, Gil D, Rodriguez M, Garcia-Reyes M, Martinez-Carnovale L, Marrero C, Gil M, Ruiz-Rodriguez JC, Ferrer R, de Nadal M, Monreal M, Llagostera S. COVID-19 Infection in Critically Ill Patients Carries a High Risk of Venous Thrombo-embolism. Eur J Vasc Endovasc Surg. 2021 Apr;61(4):628-634. doi: 10.1016/j.ejvs.2020.12.015. Epub 2020 Dec 23. PMID 33583710
- [Background] Wu C, Liu Y, Cai X, Zhang W, Li Y, Fu C. Prevalence of Venous Thromboembolism in Critically Ill Patients With Coronavirus Disease 2019: A Meta-Analysis. Front Med (Lausanne). 2021 Apr 29;8:603558. doi: 10.3389/fmed.2021.603558. eCollection 2021. PMID 33996843
- [Derived] Marrero Eligio De La Puente CE, Flota Ruiz D, Besalduch LS, Capo XF, Sala DG, Ibars CP, Mindiolaza IB, Chiscano Camon LS, Sanmartin AR, Ruiz-Rodriguez JC, Ferrer R, Montoya SB. Systematic Ultrasound Screening for Lower Extremity Deep Vein Thrombosis in ICU Patients with Severe COVID-19: A Randomized Clinical Trial. J Intensive Care Med. 2025 Jul;40(7):739-748. doi: 10.1177/08850666251313774. Epub 2025 Jan 22. PMID 39838947